CLINICAL TRIAL: NCT06679946
Title: An Open-Label Extension Study to Assess the Safety and Efficacy of Vutrisiran in Patients With Transthyretin Amyloidosis With Cardiomyopathy (ATTR Amyloidosis With Cardiomyopathy)
Brief Title: A Study to Evaluate Vutrisiran in Patients With Transthyretin Amyloidosis With Cardiomyopathy
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-TTRSC02-007; 2024-516568-27 (EudraCT Number)
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Transthyretin Amyloidosis (ATTR) With Cardiomyopathy
Keywords: ATTR; Cardiomyopathy; Amylodosis; TTR; Transthyretin; TTR-mediated amyloidosis; Amyloidosis, Hereditary, Transthyretin-Related; RNAi therapeutic; Transthyretin amyloid cardiomyopathy; TTR cardiomyopathy; ATTR-CM; Wild-type TTR; V122I; TTR amyloidosis; Amyloidosis, Wild Type; hATTR amyloidosis with cardiomyopathy; ATTR amyloidosis with cardiomyopathy; wtATTR amyloidosis with cardiomyopathy
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Cardiomyopathies; Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vutrisiran 25 mg (Experimental): Participants will receive vutrisiran 25 mg administered subcutaneously (SC) once every 3 months (q3M).
  Interventions: Drug: Vutrisiran

INTERVENTIONS:
Drug: Vutrisiran — Vutrisiran administered SC q3M
  Other Names: ALN-TTRSC02; AMVUTTRA®

SUMMARY:
The purpose of this study is to obtain safety, efficacy, and pharmacodynamic data on the use of vutrisiran in patients with ATTR amyloidosis with cardiomyopathy who continued on extended use of vutrisiran, or switched from patisiran.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are participating in the patisiran parent studies ALN-TTR02-011 or ALN-TTR02-014 or who have completed the 24-month OLE Period in the vutrisiran parent study ALN-TTRSC02-003

Exclusion Criteria:

* Has permanently discontinued study drug administration while participating in the parent studies, ALN-TTR02-011, ALN-TTR02-014, or ALN-TTRSC02-003
* Future or current participation in another investigational device or drug study, scheduled to occur during this study
* Has other medical conditions or comorbidities which, in the opinion of the Investigator, would interfere with study compliance or data interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) | Up to 36 Months
  An AE is any untoward medical occurrence in a patient or clinical investigational subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change from Baseline in the Kansas City Cardiomyopathy Questionnaire Overall Summary (KCCQ-OS) | Baseline up to 36 Months
  The KCCQ is a 23-item self-administered questionnaire quantifying 6 domains (symptoms, physical function, quality of life, social limitation, self-efficacy, and symptom stability) and 2 summary scores (clinical and overall summary [OS]). Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Change from Baseline in New York Heart Association (NYHA) Class | Baseline up to 36 Months
  NYHA classification grades the severity of heart failure symptoms into the following stages: I (no symptoms; ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea), II (symptoms with ordinary physical activity; walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea), III (symptoms with less than ordinary physical activity; walking 1 to 2 blocks on the level and climbing more than 1 flight of stairs in normal conditions causes undue fatigue or dyspnea), IV (symptoms at rest; inability to carry on any physical activity without fatigue or dyspnea).
Change From Baseline in the Cardiac Biomarker: N-terminal Prohormone of B-type Natriuretic Peptide (NT-proBNP) | Baseline up to 36 Months
  NT-proBNP will be assessed through measurement of serum levels.
Change From Baseline in the Cardiac Biomarker: Troponin I | Baseline up to 36 Months
  Troponin I will be assessed through measurement of serum levels.
All-Cause Mortality and Recurrent Cardiovascular (CV) Events (CV Hospitalizations and Urgent Heart Failure [HF] Visits) | Up to 36 Months
  All deaths, hospitalizations and urgent HF visits will be recorded throughout the study as part of SAE and AE monitoring
Change from baseline in serum TTR level | Baseline, Month 6 and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (64):
- United States (22):
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, Beverly Hills, California
  - Clinical Trial Site, La Jolla, California
  - Clinical Trial Site, Stanford, California
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Glenview, Illinois
  - Clinical Trial Site, Indianapolis, Indiana
  - Clinical Trial Site, Kansas City, Kansas
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Omaha, Nebraska
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Cleveland, Ohio
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Salt Lake City, Utah
- Argentina (2):
  - Clinical Trial Site, Rosario, S
  - Clinical Trial Site, Córdoba, X
- Clinical Trial Site, Vienna, Austria
- Belgium (4):
  - Clinical Trial Site, Liège, LIE
  - Clinical Trial Site, Hasselt, LIM
  - Clinical Trial Site, Aalst, OVL
  - Clinical Trial Site, Roeselare, WVL
- Brazil (3):
  - Clinical Trial Site, Rio de Janeiro, Rio de Janeiro
  - Clinical Trial Site, Ribeirão Preto, São Paulo
  - Clinical Trial Site, São Paulo, São Paulo
- Clinical Trial Site, Prague, Czechia
- Denmark (3):
  - Clinical Trial Site, Aarhus N
  - Clinical Trial Site, København Ø
  - Clinical Trial Site, Odense C
- France (5):
  - Clinical Trial Site, Créteil, Val-de-Marne
  - Clinical Trial Site, Marseille
  - Clinical Trial Site, Paris
  - Clinical Trial Site, Rennes
  - Clinical Trial Site, Toulouse
- Italy (3):
  - Clinical Trial Site, Bologna, Emilia-Romagna
  - Clinical Trial Site, Florence
  - Clinical Trial Site, Pavia
- Netherlands (3):
  - Clinical Trial Site, Maastricht, LI
  - Clinical Trial Site, Groningen
  - Clinical Trial Site, Utrecht
- Clinical Trial Site, Oslo, Norway
- Portugal (3):
  - Clinical Trial Site, Creixomil
  - Clinical Trial Site, Lisbon
  - Clinical Trial Site, Viseu
- Spain (3):
  - Clinical Trial Site, Barcelona, B
  - Clinical Trial Site, L'Hospitalet de Llobregat, B
  - Clinical Trial Site, Madrid
- Sweden (3):
  - Clinical Trial Site, Gothenburg
  - Clinical Trial Site, Solna
  - Clinical Trial Site, Umeå
- Clinical Trial Site, Taipei, Taiwan
- United Kingdom (6):
  - Clinical Trial Site, Birmingham, BIR
  - Clinical Trial Site, London, LND
  - Clinical Trial Site, Hexham, NBL
  - Clinical Trial Site, Bellshill
  - Clinical Trial Site, Cardiff
  - Clinical Trial Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Access to data may be declined where there is likelihood a patient could be identified or other feasibility issue, where there is a potential conflict of interest, a planned business activities or an actual or potential competitive risk. Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Timeframes for data access may vary and can take up to 6 months or more.
  Requests for access to data can be submitted via the website www.vivli.org. Questions can also be directed to datasharing@alnylam.com.

REFERENCES:
- [Result] Fontana M, Berk JL, Gillmore JD, Witteles RM, Grogan M, Drachman B, Damy T, Garcia-Pavia P, Taubel J, Solomon SD, Sheikh FH, Tahara N, Gonzalez-Costello J, Tsujita K, Morbach C, Pozsonyi Z, Petrie MC, Delgado D, Van der Meer P, Jabbour A, Bondue A, Kim D, Azevedo O, Hvitfeldt Poulsen S, Yilmaz A, Jankowska EA, Algalarrondo V, Slugg A, Garg PP, Boyle KL, Yureneva E, Silliman N, Yang L, Chen J, Eraly SA, Vest J, Maurer MS; HELIOS-B Trial Investigators. Vutrisiran in Patients with Transthyretin Amyloidosis with Cardiomyopathy. N Engl J Med. 2025 Jan 2;392(1):33-44. doi: 10.1056/NEJMoa2409134. Epub 2024 Aug 30. PMID 39213194
- See also: ALN-TTR02-011 ClinicalTrials.gov posting — https://clinicaltrials.gov/study/NCT03997383?term=ALN-TTR02-%20011&rank=1
- See also: ALN-TTR02-014 ClinicalTrials.gov posting — https://clinicaltrials.gov/study/NCT05505838?term=ALN-TTR02-%20014&rank=1
- See also: ALN-TTRSC02-003 ClinicalTrials.gov posting — https://clinicaltrials.gov/study/NCT04153149?term=ALN-TTRSC02-%20003&rank=1